CLINICAL TRIAL: NCT00553319
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Mixed Amphetamine Salts (Adderall-XR) for the Treatment of Adult Attention Deficit Hyperactivity Disorder (ADHD) and Cocaine Dependence
Brief Title: Study of Adderall-XR for the Treatment of Adult Attention Deficit Hyperactivity Disorder and Cocaine Dependence
Acronym: CAMP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #5502/6569R.; R01DA023652-01 (NIH)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder; Cocaine Dependence
Keywords: ADHD; Cocaine; Treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cocaine-Related Disorders | interventions — SLI381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Adderall-XR 60 mg (Experimental): Adderall-XR 60 mg
  Interventions: Drug: Adderall-XR
- Adderall-XR 80 mg (Experimental): Adderall-XR 80 mg
  Interventions: Drug: Adderall-XR

INTERVENTIONS:
Drug: Placebo — Placebo group
  Arms: Placebo
Drug: Adderall-XR — Adderall-XR 60mg/day
  Other Names: Extended-Release Mixed Amphetamine Salts (Adderall-XR)
  Arms: Adderall-XR 60 mg
Drug: Adderall-XR — Adderall-XR 80mg/day
  Other Names: Extended-Release Mixed Amphetamine Salts (Adderall-XR)
  Arms: Adderall-XR 80 mg

SUMMARY:
The proposed protocol is a 3 group double-blind, placebo-controlled outpatient study of the safety and efficacy of Adderall-XR (ER-MAS) in the treatment of comorbid ADHD and cocaine dependence. Since this medication has independently shown promise in helping with ADHD and cocaine abuse, we are proposing that it may be successful in the treatment of comorbid ADHD and cocaine abuse. We plan to enroll 75 subjects in a 14-week trial. The primary objectives of the study are to determine the efficacy of ER-MAS in promoting cocaine abstinence and improvement in ADHD symptomology among cocaine-dependent patients with comorbid ADHD.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the efficacy of ER-MAS in promoting cocaine abstinence and ADHD improvement among comorbid ADHD and cocaine-dependent patients.

Primary Hypothesis: benzoylecgonine positive urine screens will decrease with greatest to least reductions from 80mg>60mg>PBO (placebo).

Hypothesis 2: ADHD-Rating Scale will decrease with greatest to least reductions from 80mg>60mg>PBO.

Specific Aim 2: To determine the effect of ER-MAS on improving general functioning and impulsivity among comorbid ADHD and cocaine-dependent patients.

Hypothesis 4: There will be greater improved CGI (clinical global impression scale) scores in participants receiving d-AMPH (d-amphetamine) compared to PBO.

Hypothesis 5: ER-MAS will decrease impulsivity as measured by several self-report (Barratts Impulsivity Scale) and behavioral measures (Card Sort, IMT (immediate memory task), DMT (delayed memory task), BART) compared to PBO.

This 14-week, three arm (two medication doses versus PBO), prospective, parallel groups, randomized PBO-controlled trial with a lead-in as well as medication run-up and run down weeks, will provide clear data on efficacy and safety for definitive Phase III trials, which if successful will lead to improved treatment for A-ADHD/S-SUD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18-60 who meet DSM-IV criteria for current cocaine dependence and adult ADHD (DSM-IV-TR).
2. Used cocaine at least four days in the past month
3. Must have a Body Mass Index (BMI) > 18 kg/m2
4. Alcohol Breathalyzer (BraC) at consent of < 0.04%
5. Individuals must be capable of giving informed consent and capable of complying with study procedures.
6. Women of child bearing age will be included in the study provided that they are not pregnant, based on the results of a blood pregnancy test drawn at the time of screening. They must also agree to use a method of contraception with proven efficacy and agree not to become pregnant during the study. To confirm this, blood pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study medication. If a woman becomes pregnant, the study medication will be discontinued.

Exclusion Criteria:

1. Meets DSM-IV-TR criteria for bipolar disorder, schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse.
2. Individuals with any current Axis I psychiatric disorder as defined by DSM-IV-TR supported by the SCID-I/P that in the investigator's judgment are unstable or would be disrupted by study medication or are likely to require pharmacotherapy during the study period.
3. Individuals with current major depressive disorder.However,individuals who are currently stable on a psychotropic medication for three months with a HAM-D <14 may be included.
4. Individuals physiologically dependent on any other drugs (excluding nicotine or cannabis) which require medical intervention.
5. Individuals with current suicidal risk.
6. Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG, cardiac symptoms, fainting, open-heart surgery and/or arrhythmia, and family history of ventricular tachycardia/sudden death.
7. Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension (SBP > 140, DBP> 90, or HR > 100 when sitting quietly), acute hepatitis (patients with chronic mildly elevated transaminases < 3x upper limit of normal are acceptable), or uncontrolled diabetes.
8. Individuals with a history of seizures
9. History of allergic reaction to candidate medication (amphetamine and/or ER-MAS).
10. Women who are pregnant or nursing.
11. History of failure to respond to a previous adequate trial of the candidate medication for cocaine dependence
12. Individuals who are legally mandated (e.g., to avoid incarceration, monetary or other penalties, etc.) to participate in substance abuse treatment program
13. History of glaucoma
14. Individuals who report use of MAOI within 14 days of study start

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2007-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, MD, Principal Investigator — Columbia University; John Grabowski, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Ambulatory Research Center/Fairview University Psychiatry Dept, Minneapolis, Minnesota
  - STARS, New York, New York

REFERENCES:
- [Derived] Levin FR, Mariani JJ, Specker S, Mooney M, Mahony A, Brooks DJ, Babb D, Bai Y, Eberly LE, Nunes EV, Grabowski J. Extended-Release Mixed Amphetamine Salts vs Placebo for Comorbid Adult Attention-Deficit/Hyperactivity Disorder and Cocaine Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Jun;72(6):593-602. doi: 10.1001/jamapsychiatry.2015.41. PMID 25887096
- See also: Substance Treatment and Research Service of Columbia University — http://www.stars.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of a one week single blind placebo run-in prior to group assignment. 139 participants were enrolled and 126 were randomized following the placebo run-up
Period: Overall Study
Arm/Group | Placebo | Adderall-XR 60 mg | Adderall-XR 80 mg
Started | 43 | 40 | 43
Completed | 29 | 30 | 34
Not Completed | 14 | 10 | 9
Not completed — Lost to Follow-up | 10 | 9 | 5
Not completed — wanted treatment elsewhere | 2 | 1 | 1
Not completed — non-compliance | 0 | 0 | 2
Not completed — incarceration | 1 | 0 | 0
Not completed — moved | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Description of 126 participants randomized to study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adderall-XR 60 mg | Adderall-XR 80 mg | Total
Number analyzed (Participants) | 43 | 40 | 43 | 126
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 39.3 (7.4) | 43.9 (7.5) | 38.4 (8.6) | 40.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 20
  Male | 38 | 33 | 35 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 5
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 9 | 6 | 22
  White | 24 | 21 | 27 | 72
  More than one race | 10 | 8 | 8 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Days of cocaine use (prior 28 days) [Mean (Standard Deviation); unit: DAYS] | 11.3 (7.5) | 12.4 (7.8) | 11.3 (7.0) | 11.7 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Last Three Weeks of Cocaine Abstinence Based on Urine Toxicology Results and Self Reported Use
Description: Each week after randomization was scored dichotomously as cocaine positive or negative. Cocaine use was positive if any urine or self-report was positive. Cocaine use was negative if all urines (BE <300 ng/ml) and all self-report were negative. Weeks with no urine or no self-report were designated missing.
Time Frame: weekly for 14 weeks of trial or for length of participation
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adderall-XR 60 mg | Adderall-XR 80 mg
Number analyzed (Participants) | 43 | 40 | 43
percentage of participants | 7 | 18 | 30

2. Primary Outcome: ADHD Symptoms Based on ADHD Rating Scale
Description: The proportion of subjects exhibiting >30% reduction of AISRS score at last enrollment week compared to week 0
Time Frame: measured once per week for 14 weeks or length of study participation
Measure: Number; unit: participants
Arm/Group | Placebo | Adderall-XR 60 mg | Adderall-XR 80 mg
Number analyzed (Participants) | 43 | 40 | 43
participants | 17 | 30 | 25

ADVERSE EVENTS:
Time Frame: During 14 weeks of trial or length of study participation
Arm/Group | Placebo | Adderall-XR 60 mg | Adderall-XR 80 mg
Serious Adverse Events (participants affected / at risk) | 2/43 | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 8/43 | 19/40 | 19/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Adderall-XR 60 mg (N=40) | Adderall-XR 80 mg (N=43)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
rape (General disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Adderall-XR 60 mg (N=40) | Adderall-XR 80 mg (N=43)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (6) | 7 (7)
Insomnia (General disorders) | 1 (1) | 5 (5) | 7 (7)
Dry Mouth (General disorders) | 0 (0) | 7 (7) | 5 (5)
Decreased Appetite (General disorders) | 1 (1) | 5 (5) | 4 (4)
Fidgety/Jittery (General disorders) | 1 (1) | 2 (2) | 3 (3)
headache (General disorders) | 3 (3) | 2 (2) | 0 (0)
Racing heart (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The dropout rate was relatively low, however, there were dropouts, and this does introduce uncertainly into the outcome assessment. Since all patients received CBT we cannot conclude whether CBT is necessary to derive benefit from the medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes